CLINICAL TRIAL: NCT00164203
Title: The Feelings Club: Evaluating a School-based Intervention for Children at Risk for Depression and Anxiety Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Dr.Katarina Manassis, CAMH
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CBT_FC
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): School-based, 12-session protocol, weekly
  Interventions: Behavioral: Cognitive Behavioral Therapy; Behavioral: School-based CBT
- activity control condition (Active Comparator): Structured games and activities, weekly for 12 weeks
  Interventions: Behavioral: activity control condition

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — 12-session, weekly, school-based protocol based on cognitive restructuring, tailored to children Grades 3 to 6; comparison with activity control condition of equal duration.
  Arms: Cognitive Behavioral Therapy
Behavioral: School-based CBT — 12 sessions, weekly
  Arms: Cognitive Behavioral Therapy
Behavioral: activity control condition — weekly games & activities x 12 weeks
  Arms: activity control condition

SUMMARY:
Anxiety and mood disorders are among the most prevalent mental health problems in childhood. They have severe long-term morbidity, and associated academic and social impairment.

Building on the investigators' experience with outcome evaluation in clinically anxious or depressed children, they propose to evaluate within the school system a cognitive behavioral therapy (CBT) intervention for children in grades 3 to 6 with elevated symptoms of anxiety or depression on standardized questionnaires.

The participant's outcomes will be compared with those of similar children randomly assigned to an activity control group.

Hypothesis 1a): Children in the intervention condition will show greater symptom reduction relative to children in the control condition (primary outcome: anxiety symptoms).

Hypothesis 1b): Children in the intervention condition will show fewer symptoms during follow-up relative to children in the control condition.

Hypothesis 2: Children with anxious or depressive symptoms treated in the school setting using CBT have a lower risk of developing internalizing disorders within 1 year of treatment than children in a control condition.

Hypothesis 3: Self-esteem, anxiety and depression-related impairment, and academic functioning will improve more in intervention participants than in controls.

Hypothesis 4: School characteristics, child age, and attitudes of participating personnel are predictive of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Children with t-score elevations > 60 on either the total score or at least 4 subscales of either instrument will be considered eligible for the study.

Exclusion Criteria:

* Children will be excluded if they already meet criteria for disorders on the Anxiety Disorders Interview Schedule (ADIS), are unable to complete the inventories due to intellectual impairment or weak English skills (limiting the benefits of cognitive behavioral therapy), or if they are already engaged in ongoing psychiatric or psychological treatment that could confound study intervention effects.
* Children with elevated 'externalizing' scores on the Child Behavior Checklist (CBCL) (t-score > 60) will also be excluded, as they are often difficult to manage in CBT groups, and may obtain more benefit from other interventions.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2005-04; Primary Completion 2007-12 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Children's Depression Inventory, Multi Anxiety Scale for children, Harter Inventory and Social Skills Rating Scale | pre/post intervention; 1-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Manassis, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada